CLINICAL TRIAL: NCT05089500
Title: A Prospective Multicenter Clinical Study of a Soft Endoscopic Treatment Protocol for Internal Hemorrhoid at Degree I-Ⅲ.
Brief Title: The Two Treatment Methods Compared the Sclerosing Agent Injection and the Rubber Wrapping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Zhejiang University (Other); The First Affiliated Hospital of Nanchang University (Other); Army Military Medical University Southwestern Hospital (Unknown); Shanxi Provincial Coal Central Hospital (Unknown); Hubei Hospital of Traditional Chinese Medicine (Other); Wuhan Puren Hospital (Other); Wuhan Tianyou Hospital (Unknown); Hanyang University (Other); Enshi State Central Hospital (Unknown); Yichang Central People's Hospital (Other); Central Hospital of Xiaogan (Other); Xiaogan City First People's Hospital (Unknown); Fuyang City Second People's Hospital (Unknown); Chibi City People's Hospital (Unknown)
Responsible Party: Principal Investigator, ChenMingkai, Professor, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2021-K131
Record Dates: First submitted 2021-10-14; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Hemorrhoid; Hemorrhoids; Hemorrhoids Internal; Hemorrhoid Prolapse; Hemorrhoid Bleeding; Hemorrhoid Pain
Keywords: Endoscopic injection sclerotherapy; Endoscopic Band Ligation; Hemorrhoids; Hemorrhoid; Soft Endoscopy
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic injection sclerotherapy (Experimental)
  Interventions: Other: Endoscopic injection sclerotherapy
- Endoscopic Band Ligation (Experimental)
  Interventions: Other: Endoscopic Band Ligation

INTERVENTIONS:
Other: Endoscopic injection sclerotherapy — Patients were randomized assigned to the EIS group, preparing disposable endoscopic injections and sclerosing which were routinely administered with 1% polycinol.The transparent cap was fixed at the front end of the endoscope in inverted or orthofield of view.The stiffening agent or foam stiffer added to Meilan was injected with a disposable injection needle at 4-6 points at the oral end near the dentate line. Each point contained 0.2-1ml, and stopped after the hemorrhoid nucleus changed color. If necessary, a transparent cap was pressed to stop the bleeding to distribute the stiffening agent evenly.
  Other Names: EIS
  Arms: Endoscopic injection sclerotherapy
Other: Endoscopic Band Ligation — Patients were randomized assigned to the EBL group and were to be prepared before surgery.After the socket is mounted at the inner lens end, the socket is obviously tied at 1-2cm hemorrhoids at the mouth above the dentate line, usually 2-4 rings.With mucosal prolapse, pericyclic multiple dislocation ligation can be performed 2-3cm above the obvious prolapse.
  Other Names: EBL
  Arms: Endoscopic Band Ligation

SUMMARY:
This study is a prospective, multicentre, and randomized-controlled clinical study.The researchers wanted to explore the optimal treatment regimen for soft hemorrhoid within I-Ⅲ degrees by evaluating and comparing the effectiveness, safety and cost effect ratio of sclerosing injection and rubber lap ligation in patients with different internal hemorrhoid scores

DETAILED DESCRIPTION:
From November 2021 to July 2022, patients with internal hemorrhoids seeking treatment were enrolled according to the following criteria:

1. Age 18 to 75, men and women;
2. Patients with clinical symptoms of degree I-Ⅲ internal hemorrhoids confirmed after medical history collection, clinical examination or colonoscopy;
3. The patient was willing to receive minimally invasive treatment for internal hemorrhoids and sign informed consent by himself or his legal agent.

Exclusion criteria are as follows:

1. age <18 or> 75;
2. External hemorrhoids or mixed hemorrhoids;
3. Ⅳ degree of hemorrhoid
4. Unsymptomatic internal hemorrhoids;
5. Internal hemorrhoids were combined with complications such as chimerism, thrombosis, ulceration, or infection;
6. Poor basic conditions can not tolerate endoscopic treatment, such as serious cardiovascular and cerebrovascular diseases, respiratory dysfunction, liver and kidney failure, mental disorders, etc.;
7. There are other serious diseases involving the rectum and anus, such as anal fistula, perianal infection, anal stenosis, inflammatory bowel disease activity period, colorectal tumors, etc.;
8. Patients with severe coagulation dysfunction or long-term oral anticoagulant drugs or antiplatelet aggregation drugs without withdrawal;
9. Women in pregnancy or puerperium;
10. Sclerotic with allergy patient , such as polycininol, etc;
11. Previous history of endoscopic treatment of hemorrhoid disease, surgical history or other low rectal and anal surgery history;
12. The patient was unwilling to receive endoscopic treatment for internal hemorrhoids, and himself or his legal agent refused to sign the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75, men and women;
2. Patients with clinical symptoms of degree I-Ⅲ internal hemorrhoids confirmed after medical history collection, clinical examination or colonoscopy;
3. The patient was willing to receive minimally invasive treatment for internal hemorrhoids and sign informed consent by himself or his legal agent.

Exclusion Criteria:

1. Age <18 or age> 75;
2. External hemorrhoids or mixed hemorrhoids;
3. degree Ⅳ internal hemorrhoids
4. Unsymptomatic internal hemorrhoids
5. Internal hemorrhoids were combined with complications such as chimerism, thrombosis, ulceration, or infection；
6. Poor basic conditions can not tolerate endoscopic treatment, such as serious cardiovascular and cerebrovascular diseases, respiratory dysfunction, liver and kidney failure, mental disorders, etc.;
7. There are other serious diseases involving the rectum and anus, such as anal fistula, perianal infection, anal stenosis, inflammatory bowel disease activity period, colorectal tumors, etc.;
8. Patients with severe coagulation dysfunction or long-term oral anticoagulant drugs or antiplatelet aggregation drugs without withdrawal;
9. Women in pregnancy or puerperium;
10. Hardening agent allergy patients, such as polycininol, etc;
11. Previous history of endoscopic treatment of hemorrhoid disease, surgical history or other low rectal and anal surgery history;
12. The patient was unwilling to receive endoscopic treatment for internal hemorrhoids, and himself or his legal agent refused to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 984 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
recurernce rate | 12 months
  After treatment, the recurrence of internal hemorrhoids symptoms (based on Goligher score and HDSS symptom score)

SECONDARY OUTCOMES:
Postoperative complications and adverse events | 12 months
  Patients from complications and serious adverse events following intervention
Surgical costs | 12 months
  Cost of treatment
Health-related QIL score | 12 months
  Assessment of patient quality of life after surgery
Patient satisfaction survey | 12 months
  Patient satisfaction evaluation of the treatment method

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, M.D, Principal Investigator — Renmin Hospital of Wuhan University
Locations (2):
- China (2):
  - Mingkai Chen, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei

REFERENCES:
- [Result] Elbetti C, Giani I, Novelli E, Fucini C, Martellucci J. The single pile classification: a new tool for the classification of haemorrhoidal disease and the comparison of treatment results. Updates Surg. 2015 Dec;67(4):421-6. doi: 10.1007/s13304-015-0333-0. Epub 2015 Nov 7. PMID 26547759
- [Result] Peery AF, Crockett SD, Barritt AS, Dellon ES, Eluri S, Gangarosa LM, Jensen ET, Lund JL, Pasricha S, Runge T, Schmidt M, Shaheen NJ, Sandler RS. Burden of Gastrointestinal, Liver, and Pancreatic Diseases in the United States. Gastroenterology. 2015 Dec;149(7):1731-1741.e3. doi: 10.1053/j.gastro.2015.08.045. Epub 2015 Aug 29. PMID 26327134
- [Result] Johanson JF, Sonnenberg A. The prevalence of hemorrhoids and chronic constipation. An epidemiologic study. Gastroenterology. 1990 Feb;98(2):380-6. doi: 10.1016/0016-5085(90)90828-o. PMID 2295392
- [Result] Cosman BC. Piles of Money: "Hemorrhoids" Are a Billion-Dollar Industry. Am J Gastroenterol. 2019 May;114(5):716-717. doi: 10.14309/ajg.0000000000000234. PMID 30998519
- [Result] van Tol RR, Kleijnen J, Watson AJM, Jongen J, Altomare DF, Qvist N, Higuero T, Muris JWM, Breukink SO. European Society of ColoProctology: guideline for haemorrhoidal disease. Colorectal Dis. 2020 Jun;22(6):650-662. doi: 10.1111/codi.14975. Epub 2020 Feb 17. PMID 32067353
- [Result] Higuero T, Abramowitz L, Castinel A, Fathallah N, Hemery P, Laclotte Duhoux C, Pigot F, Pillant-Le Moult H, Senejoux A, Siproudhis L, Staumont G, Suduca JM, Vinson-Bonnet B. Guidelines for the treatment of hemorrhoids (short report). J Visc Surg. 2016 Jun;153(3):213-8. doi: 10.1016/j.jviscsurg.2016.03.004. Epub 2016 May 18. PMID 27209079
- [Result] Davis BR, Lee-Kong SA, Migaly J, Feingold DL, Steele SR. The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Management of Hemorrhoids. Dis Colon Rectum. 2018 Mar;61(3):284-292. doi: 10.1097/DCR.0000000000001030. No abstract available. PMID 29420423
- [Result] Awad AE, Soliman HH, Saif SA, Darwish AM, Mosaad S, Elfert AA. A prospective randomised comparative study of endoscopic band ligation versus injection sclerotherapy of bleeding internal haemorrhoids in patients with liver cirrhosis. Arab J Gastroenterol. 2012 Jun;13(2):77-81. doi: 10.1016/j.ajg.2012.03.008. Epub 2012 Apr 24. PMID 22980596
- [Result] Rubbini M, Ascanelli S. Classification and guidelines of hemorrhoidal disease: Present and future. World J Gastrointest Surg. 2019 Mar 27;11(3):117-121. doi: 10.4240/wjgs.v11.i3.117. PMID 31057696
- [Result] Rorvik HD, Styr K, Ilum L, McKinstry GL, Dragesund T, Campos AH, Brandstrup B, Olaison G. Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum. 2019 Mar;62(3):333-342. doi: 10.1097/DCR.0000000000001234. PMID 30451751